CLINICAL TRIAL: NCT00500916
Title: Different Techniques for Insertion of the ProSeal Laryngeal Mask Airway in Patients With Difficult Airway
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Medical University Innsbruck, Christian Keller MD, M.Sc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UN2532
Record Dates: First submitted 2007-07-11; First posted 2007-07-13 (Estimated); Last update posted 2007-12-04 (Estimated); Status verified 2007-12

CONDITIONS: Difficult Airway; Ventilation
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: ProSeal LMA — GEB vs digital vs introducer tool

SUMMARY:
The ProSeal laryngeal mask airway (PLMA) is a new laryngeal mask device with a modified cuff to improve the seal and a drain tube to prevent aspiration and gastric insufflation. The manufacturer recommends inserting the PLMA using digital manipulation, like the Classic LMA, or with an introducer tool (IT), like the Intubating LMA. The mean (range) frequency of insertion success at the first attempt for these techniques is 84% (81-100) and 95% (90-100) respectively, with the main causes of insertion difficulty being impaction at the back of the mouth and failure of the distal cuff to reach the hypopharynx. Howarth et al described an insertion technique which overcomes these difficulties by using a gum elastic bougie (GEB) placed in the esophagus to guide the PLMA around the back of the mouth and into its correct position in the hypopharynx. Howarth et al reported no failed uses from 100 consecutive insertions. In the following study, we test the hypothesis that GEB-guided insertion is more frequently successful than the digital and IT techniques in patients with difficult airway.

ELIGIBILITY:
Inclusion Criteria:

* Female patient
* 19-70 yr
* Body mass index <35 kg/m2
* Difficult airway

Exclusion Criteria:

* < 19 yr
* Body mass index >35 kg/m2
* Risk of aspiration

Ages: 19 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Estimated)
Dates: Start 2007-03; Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Insertion success rate | 5 min

SECONDARY OUTCOMES:
Time to successful insertion | 5 min

CONTACTS AND LOCATIONS:
Overall Officials: Christian Keller, MD, M.Sc., Principal Investigator — Dept of Anesthesia and Intensive Care
Locations (1):
- Department of Anesthesia and Intensive Care, Innsbruck, Austria

REFERENCES:
- [Derived] Eschertzhuber S, Brimacombe J, Hohlrieder M, Stadlbauer KH, Keller C. Gum elastic bougie-guided insertion of the ProSeal laryngeal mask airway is superior to the digital and introducer tool techniques in patients with simulated difficult laryngoscopy using a rigid neck collar. Anesth Analg. 2008 Oct;107(4):1253-6. doi: 10.1213/ane.0b013e31817f0def. PMID 18806036